CLINICAL TRIAL: NCT02851992
Title: A Prospective Study to Evaluate Long-term Clinical Outcomes of the GTS Cementless Femoral Stem
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO.CR.H36
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GTS cementless stem (Other): Total Hip arthroplasty with GTS cementless stem (standard and lateralized) with different cup and bearing options (metal-on-polyethylene or ceramic-on-polyethylene)
  Interventions: Device: GTS cementless stem

INTERVENTIONS:
Device: GTS cementless stem — Total Hip Arthroplasty

SUMMARY:
This is a multicenter, non-controlled, prospective study. 303 subjects (GTS standard and lateralized) have been recruited. Study will be conducted in centers across Europe.

DETAILED DESCRIPTION:
The objective of this prospective clinical study is to obtain multi-center, long-term (10-year) clinical data on the new GTS® femoral stem in its standard and lateralized versions as part of Post Market Surveillance requirements.

The initial study assessment period will be 12 years; 24 months recruitment and the follow-up clinical reviews for all patients will be at 3 months, 1 year, 2 years, 3 years, 5 years, 7 years and 10 years.

ELIGIBILITY:
Inclusion Criteria:

Patients inclusion criteria for this evaluation are be in accordance with the indications of the GTS® stem and specifically

* Primary osteoarthritis or secondary coxarthritis
* Inflammation of the hip: rheumatoid arthritis, etc.
* Femoral neck fracture
* Avascular necroses of the femoral head
* Sequelae from previous operations on the hip, osteotomies, etc.
* Congenital hip dysplasia

Additional inclusion criteria include:

* 18 years of age or older
* Subjects willing to return for follow-up evaluations
* Subjects who read, understood study information and provided an informed written consent (specific local regulatory requirements)

Exclusion Criteria:

Exclusion criteria are in accordance with absolute and relative contraindications for use for GTS® stem

Absolute contraindications include:

* Local or systemic infections.
* Severe muscular, neurological or vascular deficiencies of the extremity involved
* Bone destruction or poor bone quality that is likely to affect implant stability(Paget's disease, osteoporosis, etc.)
* Concomitant disease likely to affect implant function
* Allergy to any of the components of the implant
* Patients weighing more than 110 kg

Additional exclusion criteria:

* Subjects unable to co-operate with and complete the study
* Dementia and/or inability to understand and follow instructions
* Neurological conditions affecting movement
* Patient over 18 under law supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2028-09 (Estimated)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GTS Cementless Stem
Started | 303
Completed | 41
Not Completed | 262

BASELINE CHARACTERISTICS:
Population: 303 patients were enrolled in the study, 22 were excluded due to receiving a different device (20) or a screen failure (2), and therefore also not included in the baseline demographic analysis.
Arm/Group | GTS Cementless Stem
Number analyzed (Participants) | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.98 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 131
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 94
  France | 50
  Italy | 40
  Spain | 75
  Netherlands | 22
Diagnosis [Count of Participants; unit: Participants]
  Primary Osteoarthritis | 225
  Osteonecrosis of the femoral neck | 18
  congenital dysplasia | 16
  Inflammatory joint disease | 8
  Post-traumatic arthritis | 5
  Femoral neck fracture | 3
  other | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Harris Hip Score
Description: Harris Hip Score (HHS) tests will be carried out pre-operatively and at each follow-up period.
  The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). To obtain a final score, the points are summed. The minimum and maximum values of the scale are 0-100, with a higher score indicating a better outcome. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70.
Time Frame: pre-operatively and 2 years post-operatively
Population: The HHS was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. The domains covered are pain, function, absence of deformity, and range of motion. The score has a maximum of 100 points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | GTS Cementless Stem
Number analyzed (Participants) | 280
Units on a scale
  pre-operatively | 50.36 (15.93)
  2 year post-operatively: number analyzed (Participants) | 205
  2 year post-operatively | 97.75 (6.5)

2. Secondary Outcome: Stability, Incidence of Radiolucencies Around the Prosthesis and Bone Remodeling
Description: The presence or absence of the following femoral radiographic findings were reported: subsidence of the stem, stem radiolucencies, calcar resorption, heterotopic ossification.
Time Frame: 1 year post-operatively
Population: per-protocol population (all participants with 1 year radiographic evaluation available)
Measure: Count of Participants; unit: Participants
Arm/Group | GTS Cementless Stem
Number analyzed (Participants) | 226
Participants
  Subsidence of the stem (1y): number analyzed (Participants) | 224
  Subsidence of the stem (1y) | 13
  stem radiolucencies (1y) | 4
  Calcar resorption (1y): number analyzed (Participants) | 223
  Calcar resorption (1y) | 3
  Heterotopic ossification (1y): number analyzed (Participants) | 223
  Heterotopic ossification (1y) | 8

3. Secondary Outcome: Patient Satisfaction
Description: EQ-5D quality of life score will be taken at every follow-up clinic and by postal questionnaire when patients are not attending a clinic.
  The EQ-5D is a standardized instrument widely used to measure health status. The questionnaire includes 5 questions referring to mobility, self-care, daily activities, pain/discomfort and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. Scores will be within the range of 0-1 with 1 corresponding to perfect health.
Time Frame: pre-operatively and 2 years post-operatively
Population: per-protocol population (number of subjects who completed the questionnaire were included in the analysis)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GTS Cementless Stem
Number analyzed (Participants) | 279
score on a scale
  pre-operatively | 0.41 (0.29)
  2 years post-operatively: number analyzed (Participants) | 226
  2 years post-operatively | 0.96 (0.15)

4. Secondary Outcome: Adverse Events/Complications
Description: The number of revisions/removals, device-related SAE's and deaths are listed.
Time Frame: until 2 years post-operatively
Population: Complications up to 2 years post-op
Measure: Count of Participants; unit: Participants
Arm/Group | GTS Cementless Stem
Number analyzed (Participants) | 281
Participants
  Revision | 3
  device-related SAE | 2
  death | 0

5. Secondary Outcome: Survivorship
Description: Survival of the implant based on the removal or intended removal of the device. The percentage of patients that still have the implant 2 years post-operative is presented here.
Time Frame: at 2 years post-op
Population: per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | GTS Cementless Stem
Number analyzed (Participants) | 281
Participants | 278

ADVERSE EVENTS:
Time Frame: up to 2 years
Description: Adverse Events are reported via a complication case report form completed by the Investigator
Arm/Group | GTS Cementless Stem
All-Cause Mortality (participants affected / at risk) | 0/281
Serious Adverse Events (participants affected / at risk) | 11/281
Other Adverse Events (participants affected / at risk) | 32/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTS Cementless Stem (N=281)
Other hip related, Cupule conflict /psoas, cup too wide (Injury, poisoning and procedural complications) | 1
Fall of patient resulting in revision (Injury, poisoning and procedural complications) | 2 — Revision of the stem
Dislocation, 2/ DISLOCATION ON 06/26/15 (Injury, poisoning and procedural complications) | 1
Other hip related, psoas tendonitis (Injury, poisoning and procedural complications) | 1
Acetabular implant failure (Injury, poisoning and procedural complications) | 1
Other hip related, left iliac fracture due to fall (Injury, poisoning and procedural complications) | 1
Dislocation (Injury, poisoning and procedural complications) | 1
Femoral implant failure and fracture of femoral shaft (Injury, poisoning and procedural complications) | 1
Other general complication and Thrombophlebitis of the calf (General disorders) | 1
Other general complication (General disorders) | 1
Revision of cup & liner due to instability (Injury, poisoning and procedural complications) | 1 — Revision of cup&liner
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTS Cementless Stem (N=281)
Withdrawn, Conflict with The Patient / Trial / Stop of Follow-Up (Social circumstances) | 1
Instability (Injury, poisoning and procedural complications) | 1
LTF (Social circumstances) | 1
Withdrawn, not willing to return (Social circumstances) | 7
Other hip related, bursitis trochanterica (General disorders) | 1
Dislocation (Injury, poisoning and procedural complications) | 1
Other hip related, the patient doesn't execute functional kine (Injury, poisoning and procedural complications) | 1
Fracture of femoral neck (Injury, poisoning and procedural complications) | 1
Haemorrhage (Cardiac disorders) | 1 — linked to an overdose of anticoagulant, slower and long rehabilitation but no consequences
Other general complication, results and scores affected by knee pathology (General disorders) | 1
Femoral implant fracture (Injury, poisoning and procedural complications) | 1
Other general complication, total hip replacement (General disorders) | 1
Other general complication, total knee replacement (General disorders) | 1
Other general complication, Gastroesophageal reflux disease (General disorders) | 1
Superficial infection (Infections and infestations) | 1
Nerve injury, dropfoot left (Nervous system disorders) | 1
Other general complication, coxarthrosis contralateral hip (General disorders) | 1
Other general complication, coxarthrosis contralateral (General disorders) | 1
Other general complications (General disorders) | 1
Nerve injury, paralysis of the extra popliteal sciatic nerve (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT02851992/Prot_SAP_000.pdf